CLINICAL TRIAL: NCT07203872
Title: Adjunctive Inflammation-resolution Therapy in Minimally-invasive Treatment of Deep Periodontal Intrabony Defect: a Pilot Randomised Controlled Trial
Brief Title: Inflammation-resolution Therapy in MINST of Periodontal Intrabony Defect: a Pilot Randomised Controlled Trial
Acronym: AIRTIM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 343438
Record Dates: First submitted 2025-09-17; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Periodontal Diseases; Periodontitis
Keywords: MINST; non-surgical; mouthwash
MeSH Terms: conditions — Periodontal Diseases; Periodontitis

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MINST + test adjunctive anti-inflammatory mouthwash (Experimental): Patients being treated with MINST non-surgical therapy with an adjunctive test mouthwash (IsoDent Paro Strong)
  Interventions: Device: IsoDent Paro Strong (Isodent Ltd. Valtakatu 4 D, 96100 Rovaniemi, Finland) mouthwash
- MINST + placebo mouthwash (Placebo Comparator): Patients being treated with MINST non-surgical therapy with an adjunctive placebo mouthwash
  Interventions: Device: Placebo mouthwash

INTERVENTIONS:
Device: IsoDent Paro Strong (Isodent Ltd. Valtakatu 4 D, 96100 Rovaniemi, Finland) mouthwash — adjunctive anti-inflammatory mouthwash
  Arms: MINST + test adjunctive anti-inflammatory mouthwash
Device: Placebo mouthwash — Contains all the inactive ingredients as the test mouthwash without the LXA4
  Arms: MINST + placebo mouthwash

SUMMARY:
The aim of this study is to assess whether and how a mouthwash containing an ingredient that reduces inflammation in combination with a recently developed treatment is more effective at improving advanced gum disease. Advanced gum disease, also called periodontitis, is an inflammation of the gums which results in decrease in bone levels supporting teeth and can result in tooth loss. Minimally invasive non-surgical treatment (MINST) is a type of deep cleaning of teeth which involves removal of plaque beneath the gum margin and reduces inflammation. In this trial we will assess the additional benefits of combining deep cleaning (MINST) with the use of a mouthwash known to have a beneficial effect on tissue healing by helping the body to 'switch off' inflammation in periodontitis. Participants may be part of a control group, where you they be treated by MINST and provided with a placebo mouthwash The placebo mouthwash does not contain the active ingredient which reduces inflammation. Neither the participants nor the investigators can decide or be aware of which mouthwash the participants be given, as this will be determined randomly and the two mouthwash packages look the same.

The duration of the study will be over six months and will consist of a total of seven appointments. The aim of this study is to assess whether we can achieve better outcomes using this mouthwash and the healing of thegums will be assessed clinically. In addition, other parameters such as saliva samples, blood samples and plaque samples will be collected throughout the study, which allows us to examine the healing process in more detail and will help us understand how exactly the combination of MINST and the mouthwash improve healing.

DETAILED DESCRIPTION:
This is a pilot randomised controlled trial comparing patients being treated with MINST non-surgical therapy with an adjunctive test or placebo mouthwash. This will be a single centre trial in the Department of Periodontology at Guy's Dental Hospital. Patients will be recruited and treated at this centre as per the inclusion criteria. The primary outcome is PPD reduction at 6 months in test vs control group, and the secondary outcomes are CAL reduction at 6 months, changes in inflammatory/tissue degradation/repair biomarkers in saliva and GCF between baseline and 6 months post-treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 70
2. Diagnosis of periodontitis stage III-IV
3. Presence of at least 1 deep intrabony defect (both PPD and radiographic defects >6mm)
4. Full-mouth dichotomous plaque score>30%
5. Willing to voluntarily sign the informed consent.

Exclusion Criteria:

1. Previous periodontal treatment to the study site within 6 months
2. Use of systemic antibiotics within 3 months
3. Weekly regular use of non-steroidal anti-inflammatory drugs
4. Contributing medical history according to the examining clinician (e.g. diabetes mellitus)
5. Smoking history (current or within 5 years)
6. Allergic to any ingredient present in the products used in study.
7. Presence of systemic diseases, which affects bone and/or connective tissue metabolism
8. Concurrent participation in other clinical studies.
9. Pregnant or breastfeeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Probing pocket depth | 6 months
  Measure of depth of periodontal pocket taken with periodontal probe (in mm)

SECONDARY OUTCOMES:
Pocket closure | 6 months
  Reduction of pocket below 5 mm
Clinical attachment level | 6 months
  Measure of periodontal attachment level taken with periodontal probe (in mm) (sum of pocket depth and gingival recession)
Patient-related outcome measures | 6 months
  OHIP-14 score recorded by patients in OHIP-14 questionnaire
Composite outcome | 6 months
  Combination of reduction of pocket depth<5mm and clinical attachment level gain of at least 3 mm (baseline- 3 months)
Changes in biomarkers | day 1, day 7, 1 month, 3 months, 6 months
  Changes in levels of mcirobial, inflammatory and host-response biomarkers in gingival crevicular fluid, subgingival plaque, saliva and blood at different points after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Oral Clinical Research Unit (OCRU) at King's College London (KCL), London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Van Dyke TE, Sima C. Understanding resolution of inflammation in periodontal diseases: Is chronic inflammatory periodontitis a failure to resolve? Periodontol 2000. 2020 Feb;82(1):205-213. doi: 10.1111/prd.12317. PMID 31850636
- [Background] Serhan CN, Chiang N. Resolution phase lipid mediators of inflammation: agonists of resolution. Curr Opin Pharmacol. 2013 Aug;13(4):632-40. doi: 10.1016/j.coph.2013.05.012. Epub 2013 Jun 6. PMID 23747022
- [Background] Nibali L, Pometti D, Chen TT, Tu YK. Minimally invasive non-surgical approach for the treatment of periodontal intrabony defects: a retrospective analysis. J Clin Periodontol. 2015 Sep;42(9):853-859. doi: 10.1111/jcpe.12443. Epub 2015 Sep 29. PMID 26257238